CLINICAL TRIAL: NCT02387762
Title: A Phase 2a, 4-Week, Double-Blind, Proof-of-Concept Efficacy and Safety Study of ACP-196 Versus Placebo in Subjects With Active Rheumatoid Arthritis on Background Methotrexate
Brief Title: ACP-196 Versus Placebo in Subjects With Rheumatoid Arthritis on Background Methotrexate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Acerta Pharma BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACE-RA-001
Record Dates: First submitted 2015-03-01; First posted 2015-03-13 (Estimated); Results first posted 2019-03-26 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Acalabrutinib
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — acalabrutinib; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ACP-196 + Methotrexate (Experimental): Oral acalabrutinib 15 mg QD plus a stable dose of methotrexate (MTX) between 7.5 mg and 25 mg per week
  Interventions: Drug: acalabrutinib
- Placebo + Methotrexate (Placebo Comparator): Oral placebo QD plus a stable dose of MTX between 7.5 mg and 25 mg per week
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: acalabrutinib
  Other Names: methotrexate
  Arms: ACP-196 + Methotrexate
Drug: Placebo
  Other Names: methotrexate
  Arms: Placebo + Methotrexate

SUMMARY:
This study is evaluating the safety, pharmacokinetics (PK), pharmacodynamics (PD) and efficacy of ACP-196 in subjects with Rheumatoid Arthritis on background Methotrexate.

DETAILED DESCRIPTION:
A multicenter, randomized, double-blind, placebo-controlled, parallel-group clinical trial. The on-treatment period is 4 weeks with weekly visits to the clinic, followed by a 4-week safety follow-up period after the last dose of ACP-196/placebo. The study was to evaluate the safety, PK, PD, and efficacy of ACP-196 in subjects with Rheumatoid Arthritis on background Methotrexate

ELIGIBILITY:
Main Inclusion Criteria:

* Diagnosis of RA according to the 2010 ACR/EULAR Classification Criteria .
* Must be on a stable MTX dose (7.5 to 25 mg/week)
* Subjects must be able to read and understand the consent form, complete the study-related procedures, and communicate with the study staff.
* Are willing and able to adhere to the study visit schedule, and understand and comply with other protocol requirements.

Main Exclusion Criteria:

* Prior malignancy, except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer from which the subject has been disease free for ≥ 5 years.
* A life-threatening illness, medical condition or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of ACP-196, or put the study outcomes at undue risk.
* Subjects who have taken any investigational drug within the previous 30 days before randomization.
* Use of all other synthetic disease-modifying antirheumatic drugs (DMARDS) such as but not limited to leflunomide, azathioprine, cyclosporine, penicillamine or gold salts within 8 weeks of randomization.
* Use of etanercept, anakinra, tofacitinib within 4 weeks of randomization.
* Use of abatacept, humira, infliximab, or tocilizumab within 8 weeks of randomization.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-04; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Acerta Clinical Trials, Study Director — Acerta Pharma, LLC
Locations (17):
- United States (17):
  - Pinnacle Research Group, Anniston, Alabama
  - Achieve Clinical Research, Birmingham, Alabama
  - Advanced Arthritis Care and Research, Scottsdale, Arizona
  - TriWest Research Associates, LLC, El Cajon, California
  - Neuropsychiatric Research Center of Orange County, Orange, California
  - Pacific Arthritis Center Medical Group, Santa Monica, California
  - Inland Rheumatology and Osteoporosis Medical Group, Inc, Upland, California
  - San Marcus Research Clinic, Inc., Hialeah, Florida
  - Suncoast Clinical Research, Inc., New Port Richey, Florida
  - Suncoast Clinical Research, New Port Richey, Florida
  - The Arthritis Center, Palm Harbor, Florida
  - Office of George Timothy Kelly, MD, Las Vegas, Nevada
  - PMG Research of Salisbury, Salisbury, North Carolina
  - Health Research of Oklahoma, Oklahoma City, Oklahoma
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Ramesh C. Gupta, MD, Memphis, Tennessee
  - Clear Lake Regional Medical Center, Webster, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ACP-196 + Methotrexate | Placebo + Methotrexate
Started | 16 | 15
Completed | 15 | 15
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population, which included all randomized subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | ACP-196 + Methotrexate | Placebo + Methotrexate | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 12 | 22
  >=65 years | 6 | 3 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (7.21) | 56.8 (7.92) | 59.1 (7.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 27
  Male | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 2 | 3 | 5
  White | 14 | 10 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 15 | 31
DAS28-CRP at baseline [Mean (Standard Deviation); unit: Scores on Scale] — Using the scores on the scale, measure disease activity score from the DAS28 scale and results from the C-reactive protein at baseline.
  Scores on Scale | 6.29 (1.242) | 6.29 (1.220) | 6.29 (1.211)
Duration of rheumatoid arthritis since initial diagnosis [Mean (Standard Deviation); unit: years] — To measure duration of rheumatoid arthritis since initial diagnosis at baseline
  years | 10.3 (7.52) | 7.8 (8.12) | 9.1 (7.78)
Methotrexate dosing at baseline [Mean (Standard Deviation); unit: mg/week] — To measure methotrexate exposure at baseline
  mg/week | 16.9 (6.49) | 17.7 (5.22) | 17.3 (5.82)

OUTCOME MEASURES:

1. Primary Outcome: Disease Activity Score 28-CRP (DAS28-CRP) at Week 4
Description: Disease activity score 28 - C-reactive protein (DAS28-CRP) is a score to measure disease activity in patients with rheumatoid arthritis by aggregating data of 28 joints, and is calculated by the scores on scale using the following variables: The number of swollen and tender joints, CRP level, and patient's global assessment of disease activity. The total score of the DAS28 values may range from 2.0 to 10.0 while higher values mean a higher disease activity.
Time Frame: 4 weeks
Population: Intent-to-treat population, which included all randomized subjects
Measure: Mean (Standard Deviation); unit: Scores on scale
Groups:
- ACP 196 + Methotrexate: Oral acalabrutinib 15 mg QD plus a stable dose of methotrexate (MTX) between 7.5 mg and 25 mg per week
Arm/Group | ACP 196 + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 15 | 15
Scores on scale | 5.40 (1.563) | 5.05 (1.639)

ADVERSE EVENTS:
Time Frame: From the date of the first dose of study drug up to 30 days after the date of the last dose of study drug, up to 6 months.
Description: Subjects with multiple events for a given system organ class (SOC) and preferred term (PT) were counted only once for each SOC and PT. If the same event term was reported more than once for a subject, only the event with the highest grade was included.
Arm/Group | ACP-196 + Methotrexate | Placebo + Methotrexate
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 10/16 | 6/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ACP-196 + Methotrexate (N=16) | Placebo + Methotrexate (N=15)
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 1
Full Blood Count decreased (Investigations) | 1 | 0
Blood uric acid increased (Investigations) | 0 | 1
Hypochloraemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Site and PI can publish/publicly present the results of the study only with prior written consent of Sponsor or otherwise after expiry of 12 months following completion of the study. Site and PI agree to provide 45 days written notice to Sponsor prior to submission for publication or presentation.